CLINICAL TRIAL: NCT05947084
Title: Comparison of Growth and Tolerance of Healthy Term Infants Fed Iron-Fortified Infant Formulas. A 4 Month, Prospective, Randomized, Multi Center Clinical Trial.
Brief Title: Comparison of Growth and Tolerance of Healthy Term Infants Fed Iron-Fortified Infant Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aussie Bubs, Inc. (Industry)
Collaborators: Validcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BubsGMS_2023
Record Dates: First submitted 2023-06-27; First posted 2023-07-17 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Infant Development
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: Randomization and exclusive feeding of study formulas by 14 days of age. Breastfed Cohort will be evaluated over the 16 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study infant formulas have been blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study Formula 1_365 Day Grass-Fed Cow's Milk Infant Formula (Experimental): Infant formula meets all nutrient requirements of the FDA.
  Interventions: Other: Infant Formula
- Study Formula 2_Goat Milk Infant Formula (Experimental): Infant Formula meets all nutrient requirements of the FDA.
  Interventions: Other: Infant Formula
- Study Formula 3_Cow's Milk Infant Formula void of A1-BetaCasein (Experimental): Infant Formula meets all nutrient requirements of the FDA.
  Interventions: Other: Infant Formula
- Study Formula 4_USDA Organic iron fortified infant formula (Active Comparator): Infant Formula meets all nutrient requirements of the FDA.
  Interventions: Other: Infant Formula

INTERVENTIONS:
Other: Infant Formula — Growth Monitoring Study of Infant Formula fed to Healthy Term Infants over a 16 week period

SUMMARY:
A 4 month growth monitoring study of healthy term infants fed iron fortified infant formula. Infants will be fed ad-libitum for 16 weeks and growth will be evaluated in terms of weight gain over the 16 weeks.

DETAILED DESCRIPTION:
A Growth Monitoring Study conducted according to FDA established guidelines to evaluate the test infant formulas ability to promote normal growth and development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Term Infant

Exclusion Criteria:

* Any health condition that would negatively impact infant feeding and growth.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 518 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Weight gain (g) from study entry to 16 weeks of study. | 16 weeks of Clinical Study
  Growth Monitoring Study

SECONDARY OUTCOMES:
Recumbent length gain (cm) from study entry to 16 weeks of study. | 16 weeks of Clinical Study
  Growth Monitoring Study
Head Circumference gain (cm) from study entry to 16 weeks of study | 16 weeks of Clinical Study
  Growth Monitoring Study
Tolerance of study formulas over 16 weeks of study | 16 weeks of Clinical Study
  Tolerance of the infant to the study formulas will be evaluated 5 times through the use of study diaries for 3 days before each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Aqua, MD, Principal Investigator — Backtee Holdings, LLC
Locations (29):
- United States (29):
  - Velocity Clinical Research-Phoenix, Phoenix, Arizona
  - Advance Pediatric Associates, Centennial, Colorado
  - Symphony Clinical Research, Jacksonville, Florida
  - Clintheory Healthcare Miami, North Miami Beach, Florida
  - PAS Research Tampa, Tampa, Florida
  - UpTo Trials, Tampa, Florida
  - Backtee Holdings, LLC, Wellington, Florida
  - Velocity Clinical Research-Macon, Macon, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Kentucky Pediatric Research, Bardstown, Kentucky
  - Springs Medical Research, Owensboro, Kentucky
  - Magnolia Clinical Research, LLC, Lutcher, Louisiana
  - Velocity Clinical Research-Slidell, LA, Slidell, Louisiana
  - Frontier Pediatric Research, LLC, Lincoln, Nebraska
  - PAS Research Henderson, Henderson, Nevada
  - PAS Research Vegas, Las Vegas, Nevada
  - Velocity Clinical Research-Durham, Durham, North Carolina
  - Hightower Clinical-Oklahoma City, Oklahoma City, Oklahoma
  - Hightower Clinical-Shawnee, Shawnee, Oklahoma
  - Cyn3rgy, Gresham, Oregon
  - PAS Pittsburgh, Pittsburgh, Pennsylvania
  - Coastal Ped Research-Charleston, Charleston, South Carolina
  - Coastal Ped Research-Summerville, Summerville, South Carolina
  - AVIATI Healthcare & Clinical Research, Memphis, Tennessee
  - Helios Clinical Research-Burleson, Burleson, Texas
  - Helios Clinical Research-Houston, Houston, Texas
  - Prime Clinical Research, Inc, Mansfield, Texas
  - PAS Research McAllen, McAllen, Texas
  - Helios Clinical Research-Weatherford, Weatherford, Texas

IPD SHARING:
Plan to Share IPD: No